CLINICAL TRIAL: NCT04578652
Title: Fiber Supplementation and Metformin Combination Therapy in Adolescents With Severe Obesity and Insulin Resistance: Interactions With the Gut Microbiome.
Brief Title: Fiber and Metformin Combination Therapy in Adolescents With Severe Obesity and Insulin Resistance
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RN. # 414120
Record Dates: First submitted 2020-09-01; First posted 2020-10-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Childhood; Insulin Resistance
Keywords: Dietary fiber; Metformin
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance | interventions — Metformin; oligofructose; Gum Arabic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and research team will be blinded to the type of intervention allocated to each arm until the end of the study. Concealment will be protected by secure, password protected website. The group not on MET (fiber alone) will receive a placebo pill. The group not on fiber will also receive a placebo, composed of the same base solution without added fibers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MET (Active Comparator): MET (850 mg po bid - standard of care) + Fiber placebo daily
  Interventions: Drug: Metformin 850 mg oral tablet bid
- FIBER (Active Comparator): Fiber supplementation [35g fiber daily] + MET placebo po bid
  Interventions: Dietary Supplement: Supplemental fiber mixture (35 g total) composed of 6g of Oligofructose + 12g of resistant maltodextrin + 12g of acacia gum + 5g of PGX.
- FIBER + MET (Experimental): Fiber supplementation [35g fiber daily] + MET 850 mg po bid
  Interventions: Drug: Metformin 850 mg oral tablet bid; Dietary Supplement: Supplemental fiber mixture (35 g total) composed of 6g of Oligofructose + 12g of resistant maltodextrin + 12g of acacia gum + 5g of PGX.

INTERVENTIONS:
Drug: Metformin 850 mg oral tablet bid — MET dose: 500 mg daily, increasing to 500 bid if tolerated after 2 weeks, then increasing again 2 weeks later to 850 mg bid (1700 mg daily).
  Arms: FIBER + MET; MET
Dietary Supplement: Supplemental fiber mixture (35 g total) composed of 6g of Oligofructose + 12g of resistant maltodextrin + 12g of acacia gum + 5g of PGX. — The first week of treatment will use 1/3 the daily treatment dose; then 2/3 dose for the second and third weeks; then the full dose thereafter, to allow time for adaptation.
  Arms: FIBER; FIBER + MET

SUMMARY:
This is a 12-month, single center, three-arm parallel design, double-blind, randomized clinical trial, to compare the effects of supplemental dietary fiber and metformin (MET) alone and in combination over 12 months on glucose metabolism (insulin resistance [IR]), inflammation and BMI in adolescents with obesity and IR, and to assess the relationship between therapeutic intervention(s) and changes in gut microbiome composition and function.

Since MET and FIBER have been shown to reduce weight and increase insulin sensitivity through distinct but overlapping mechanisms of action, our central hypothesis is that the combination of FIBER + MET will have a synergistic effect and be more effective than FIBER or MET alone in improving metabolic function (IR) and reducing BMI and inflammation in adolescents with obesity, IR and family history (FM) of T2DM.

.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-18 years
2. BMI percentile > 95% for age/sex;
3. Total weight fluctuation over past 6 months < 10%;
4. HOMA-IR > 3.16;
5. FH of T2DM (first or second-degree relative).

Exclusion Criteria:

1. Current use of insulin or diagnosis of T2DM;
2. Systolic or diastolic blood pressure (BP) > 99th percentile for age and sex;
3. Acute infectious or inflammatory condition over the preceding 1 month; hospitalization > 48 hrs;
4. History of chronic disease such as inflammatory bowel disease, chronic severe liver or kidney disease or neurologic disorders;
5. Active malignancy;
6. Concomitant use of medication/investigational drug known to affect body weight in the past year;
7. Antibiotic use in past 60 days; probiotic and/or prebiotic supplements use in the past 30 days; use of lipid-lowering and anti-inflammatory medication.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Changes in HOMA-IR | Baseline, 6, and 12 months
  Change in HOMA-IR value

SECONDARY OUTCOMES:
Changes in body weight | Baseline, 6, and 12 months
  Body weight measured in kg
Changes in body mass index (BMI) | Baseline, 6, and 12 months
  BMI percentile and z-score according to age and sex will be estimated
Changes in body composition | Baseline, 6, and 12 months
  Body density using air-displacement plethysmography will be assessed to estimate fat mass and fat-free mass.
Changes in inflammation | Baseline, 6, and 12 months
  Markers of inflammation that will be measured are: high-sensitivity C-reactive protein, interleukin, tumor necrosis factor-alpha)
Changes in metabolic function | Baseline, 6, and 12 months
  The markers of metabolic function that will be measured are: fasting glucose, lipids (total, high and low density lipoprotein cholesterol; triglycerides), and oral glucose tolerance test.
Changes in satiety hormones | Baseline, 6, and 12 months
  Markers of satiety that will be measured are: acylated ghrelin, peptide tyrosine tyrosine, GLP-1, leptin, and adiponectin.
Changes in quality of life | Baseline, 6, and 12 months
  Quality of life will be measured by the a questionnaire
Changes in perceived hunger and satiety | Baseline, 6, and 12 months
  Perceived hunger and satiety will be assessed by a questionnaire
Changes in gut microbiota composition | Baseline, 6, and 12 months
  Fecal microbiota composition will be characterized by 16S rRNA gene amplicons sequencing using taxonomic and non-taxonomic based approaches.
Changes in gut microbiome functions | Baseline, 6, and 12 months
  Fecal microbiome functions will be assessed through whole metagenomic sequencing, stool SCFAs and bile acids, and plasma metabolomics.
Changes in intestinal barrier integrity | Baseline, 6, and 12 months
  Plasma lipopolysaccharide-binding protein and fecal calprotectin will be determined as measures of gut barrier integrity

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Haqq, MD, MHS, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fahim SM, Huey SL, Palma Molina XE, Agarwal N, Ridwan P, Ji N, Kibbee M, Kuriyan R, Finkelstein JL, Mehta S. Gut microbiome-based interventions for the management of obesity in children and adolescents aged up to 19 years. Cochrane Database Syst Rev. 2025 Jul 10;7(7):CD015875. doi: 10.1002/14651858.CD015875. PMID 40637175
- [Derived] Deehan EC, Colin-Ramirez E, Triador L, Madsen KL, Prado CM, Field CJ, Ball GDC, Tan Q, Orsso C, Dinu I, Pakseresht M, Rubin D, Sharma AM, Tun H, Walter J, Newgard CB, Freemark M, Wine E, Haqq AM. Efficacy of metformin and fermentable fiber combination therapy in adolescents with severe obesity and insulin resistance: study protocol for a double-blind randomized controlled trial. Trials. 2021 Feb 17;22(1):148. doi: 10.1186/s13063-021-05060-8. PMID 33596993